CLINICAL TRIAL: NCT00105573
Title: Prevention for Infants of Low-Income Depressed Mothers
Brief Title: Interventions for Depressed Low Income Mothers and Their Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sheree Toth, Executive Director, Mt. Hope Family Center, and Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH067792 (NIH); R01MH067792 (NIH); DSIR 84-CTP
Record Dates: First submitted 2005-03-15; First posted 2005-03-16 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Depression
Keywords: Mother-Child Relations; Infant; Child Development; Poverty
MeSH Terms: conditions — Depression | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Interpersonal Psychotherapy (Experimental): Participants will receive interpersonal psychotherapy for depression.
  Interventions: Behavioral: Maternal interpersonal psychotherapy (IP)
- Interpersonal psychotherapy/child-parent psychotherapy (Experimental): Participants will receive interpersonal psychotherapy for depression plus 1 year of in-home, child-parent psychotherapy.
  Interventions: Behavioral: Maternal interpersonal psychotherapy (IP); Behavioral: Infant-parent psychotherapy
- Enhanced community standard (Active Comparator): Participants will be invited to attend informational meetings as well as be referred to local services available to people with depression.
  Interventions: Behavioral: Informational meetings plus treatment as usual

INTERVENTIONS:
Behavioral: Maternal interpersonal psychotherapy (IP) — Participants will receive 16 weekly sessions of maternal IP designed to directly treat maternal depression.
  Arms: Interpersonal Psychotherapy; Interpersonal psychotherapy/child-parent psychotherapy
Behavioral: Infant-parent psychotherapy — Participants will receive 1 year of in-home, infant-parent psychotherapy, an intervention addressing relationship difficulties between depressed mothers and their infants.
  Arms: Interpersonal psychotherapy/child-parent psychotherapy
Behavioral: Informational meetings plus treatment as usual — Participants will be invited to attend informational meetings as well as be referred to local services available to people with depression.
  Arms: Enhanced community standard

SUMMARY:
This study will compare three interventions for depressed, low income mothers and determine which is most effective in treating maternal depression and in fostering development in infants.

DETAILED DESCRIPTION:
Poorly educated, low income mothers are at high risk for becoming depressed. The effects of living in poverty and being reared by a depressed parent can be detrimental to an infant's development. Effective interventions to reduce maternal depression and strengthen the mother-infant relationships are needed.

Participants will be randomly assigned to one of three groups. Group 1 mothers will receive 16 weekly sessions of interpersonal psychotherapy (IP) designed to directly treat maternal depression. Group 1 participants will have monthly follow-up visits for 1 year. Participants in Group 2 will receive 16 weekly sessions of IP followed by 1 year of in-home, infant-parent psychotherapy, an intervention addressing relationship difficulties between depressed mothers and their infants. Group 3 mothers will be invited to attend informational meetings as well as be referred to local services available to people with depression.

All mother-child pairs will be evaluated when the child is 12, 16, 24, and 36 months of age. Evaluations will involve questionnaires, diagnostic interviews, developmental assessments, and video- and audio-taped measures.

ELIGIBILITY:
Inclusion Criteria for Mothers:

* Current diagnosis of depression
* Mother of an infant 9 to 11 months of age
* Low income, defined as less than $25,000 for a family of two or less than $31,400 for a family of three (add approximately $7,960 for each additional family member)

Exclusion Criteria for Mothers:

* Current substance abuse
* Severe mental or physical limitations that would interfere with the study

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 218 (Actual)
Dates: Start 2004-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Maternal depression | Measured when the child is 12, 16, 24, 36, and 48 months of age
Child development | Measured when the child is 12, 16, 24, 36, and 48 months of age
Infant-parent attachment | Measured when the child is 12, 16, 24, 36, and 48 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Sheree Toth, PhD, Principal Investigator — Mount Hope Family Center
Locations (1):
- Mount Hope Family Center, Rochester, New York, United States